CLINICAL TRIAL: NCT01826292
Title: The Association Between Anesthetic and Surgical Practices and Patient Length of Stay in the Post Anesthesia Care Unit
Status: Withdrawn | Type: Observational
Why Stopped: Principle Investigator was not able to proceed with the study
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 363700
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Post Anesthesia Care Unit Length of Stay
Keywords: Post anesthesia care unit length of stay

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Cross-sectional cart review
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators are conducting a retrospective, cross-sectional chart review of patients who underwent an anesthetic administered by an anesthesiologist in the University of California Davis main operating rooms and were transferred to the main post anesthesia care unit between January 1, 2012 and March 31, 2012. The investigators are excluding patients less than 18 years of age, patients transferred to the intensive care unit, and patients for whom data is not reported. Our aim is to report the incidences patient characteristics, as well as anesthetic and surgical techniques, and the associations these factors may have with the outcome of patient length of stay in the PACU.

DETAILED DESCRIPTION:
We are conducting a retrospective, cross-sectional chart review of patients who underwent an anesthetic administered by an anesthesiologist in the University of California Davis main operating rooms and were transferred to the main (Pavilion) post anesthesia care unit between January 1, 2012 and March 31, 2012. We are excluding patients less than 18-years of age, patients transferred to the intensive care unit, and patients for whom data is not reported. Charts will be reviewed and data will be collected by the primary and co-investigator(s). Analysis will consist of cross-tabulation counts across independent variables, univariate analysis (outcome variable PACU length of stay), and regression analysis (outcome variable PACU length of stay). We aim to measure patient length of stay in the post anesthesia care unit (PACU) as the outcome variable. The following patient, operative, and post operative factors will be recorded as covariates: age, gender, height, weight, American Society of Anesthesiologists physical status classification, pre-operative use of pain medication, pre-operative pain score, whether the patient is non-English speaking, history of smoking, surgical service, anesthetic time, surgical time, urgency of surgery, use of general anesthetic or monitored anesthesia care, use of regional anesthetic, regional anesthetic type, use of inhalational or total intravenous anesthetic maintenance, intraoperative use of dexmedetomidine, intraoperative use of dexamethasone, intraoperative use of ondansetron, intraoperative use of remifentanyl, intraoperative use of ketamine, total volume of crystalloid or colloid administered, intraoperative use of endotracheal tube, natural airway, or laryngeal mask airway, time of PACU arrival, initial pain score in the PACU, episode of post operative nausea or vomiting, administration of antiemetic in the PACU, post operative temperature, time of anesthesiologist sign out in the PACU, time of patient transfer from the PACU, location of transfer from PACU, preoperative placement of scopolamine patch, history of postoperative nausea and vomiting, type of surgery (including categories of major abdominal-open, orthopedic, ear nose and throat, thoracic, vascular, ophthalmology, abdominal-laparoscopic, urology, minor, neurology, and plastics), intra operative estimated blood loss, intra operative administration of the following medications: dexamethasone, antiemetics including dexamethasone, acetaminophen, ketorolac, muscle relaxant (i.e. paralytics), muscle relaxant reversal agents, and morphine equivalent dosage of opioids; intra operative volume of colloid administered, intra operative volume of blood products administered, morphine equivalent dosage of opioids administered in the post anesthesia care unit, times of admission and discharge from the post anesthesia care unit. The data will be labeled with a code that the research team can link to personal identifying information when acquired. The code sheet will be secured and kept separate from the dataset. The primary and co-investigator(s) will be the only individuals who have access to the password protected database stored on a secure server at the University of California Davis Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent an anesthetic administered by an anesthesiologist in the University of California Davis main operating rooms and were transferred to the main post anesthesia care unit between January 1, 2012 and March 31, 2012.

Exclusion Criteria:

* Patients less than 18-years of age,
* Patients transferred to the intensive care unit, and
* Patients for whom data is not reported.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent an anesthetic administered by an anesthesiologist in the University of California Davis main operating rooms and were transferred to the main post anesthesia care unit between January 1, 2012 and March 31, 2012.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Patient length of stay in the post anesthesia care unit | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Harmeet Bhullar, MD, Principal Investigator — University of California, Davis